CLINICAL TRIAL: NCT06613477
Title: Pharmacokinetics and Pharmacodynamics of Digoxin in Infants With Single Ventricle Heart Disease
Brief Title: PK/PD of Digoxin in Infants With SVHD
Acronym: Digoxin R01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Medical University of South Carolina (Other); Duke Clinical Research Institute (Other); National Center for Child Health and Development (NICHD) (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113213; 1R01HD106588-01A1 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Single-ventricle; Infant Conditions; Infant, Newborn, Diseases; Infant, Premature, Diseases
Keywords: Infants; SVD; SVHD; Single Ventricle; Digoxin; Pharmacokinetics; Pharmacodynamics; PK; PD
MeSH Terms: conditions — Univentricular Heart; Infant, Newborn, Diseases; Infant, Premature, Diseases | interventions — Digoxin

STUDY DESIGN:
Intervention Model Description: Each subject will receive population specific PK model-derived digoxin dosing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Population specific PK model-derived digoxin dosing (Experimental): Digoxin elixir will be used to dose enterally every 12 hours.
  The dosage will be determined by the protocol PK model. Dosing is to be administered based on weight, postnatal age, and estimated glomerular filtration rate
  The duration of the participation could be up to 180 days. Day 1 to S2P or Day 180 (+/- 7)
  Interventions: Drug: PK/PD Model Based Dosing of Digoxin in Infants with Single Ventricle Heart Disease

INTERVENTIONS:
Drug: PK/PD Model Based Dosing of Digoxin in Infants with Single Ventricle Heart Disease — Table 3: Digoxin dosing regimen based on optimized Cmin,ss Dose to be given twice daily (mcg/kg/dose) PNA<30 days 30 days < PNA < 180 days eGFR≤40 1.4 1.4 40<eGFR≤60 1.6 1.6 eGFR>60 1.9 2.8
  Other Names: Lanoxin

SUMMARY:
The primary participant will be an infant with single ventricle heart disease.

This is a research study to learn more about how the medication digoxin, which is routinely prescribed to infants and children with heart disease in pediatric cardiac intensive care units is processed by their bodies and how it may help their cardiac function.

The investigators will collect blood or will collect blood samples when bloodwork is checked as part of regular care ("opportunistic"). The investigators will also collect information from medical records.

Being part of this study will not change treatment plan or medications. The risks of this study include loss of confidentiality and risks associated with having blood drawn. The study team will make every effort to minimize these risks.

DETAILED DESCRIPTION:
Study design: Multi-center, prospective, open-label, opportunistic PK/PD study of digoxin.

Randomization: none Blinding /Masking: none Study intervention: Each subject will receive population specific PK model-derived digoxin dosing Duration of participant participation: up to 180 days

Table 1. PK sample collection times PK Sample # Sample window for plasma collection

1. 8 - 11.5 hours after dose / trough level on dosing Day 7 (+/- 2 days)
2. 15 minutes - 1 hour after dose on dosing Day ≥14
3. 2 - 5 hours after dose on dosing Day ≥14
4. 8 - 11.5 hours after dose / trough level on dosing Day ≥14
5. - 7* 8 - 11.5 hours after dose / trough level on any dosing Day ≥14 and ≤180 or Day of S2P

PK sampling: digoxin concentrations in plasma will be measured at a central lab using validated bioanalytical assays. Plasma samples for digoxin quantification will be drawn according to Table 1. Initial PK sample will be obtained once on dosing Day 7 (+/- 2 days). PK samples 2-4 will be obtained once on dosing day ≥14. Every effort will be made to collect samples 2-4 after the same digoxin dose. Up to 3 additional samples will be collected 8 - 11.5 hours after dosing on different dosing days ≥14 but ≤180 or day of S2P, whichever occurs first. Samples 5 - 7 will be collected on different days.

Table 2. PD sample collection times PD Sample # Sample window for plasma collection

1. Within 24 hours prior to first digoxin dose
2. Any time on dosing day 28 (+/- 7 days)
3. Any time on dosing day 112 (+/- 7 days)
4. Any time within 7 days prior to S2P

PD sampling: plasma samples for NT-proBNP and MR-proANP quantification will be collected according to Table 2.

Safety: Adverse events related to the study procedure (sample collection, blood draws and outcome assessments), adverse events related to digoxin, select events of special interest (tachyarrythmias, second and third degree atrioventricular conduction block, sinus bradycardia, need for temporary or permanent pacing, death), and serious, unexpected, suspected adverse reactions (SUSARs) related to digoxin will be captured.

Cardiac assessments: records of echocardiograms and cardiac catheterizations performed per standard of care will be collected.

This study will be conducted in accordance with current U.S. Food and Drug Administration regulations and guidelines, (or, as applicable, the European Clinical Trials Directive and associated guidelines), the International Conference on Harmonisation Guidelines on Good Clinical Practice (which incorporate the principles of the Declaration of Helsinki), as well as all other applicable national and local laws and regulations.

Scientific Rationale for Study Design This study is designed to prospectively validate the PK model-derived dosing of digoxin in infants with single ventricle CHD after S1P but before S2P. A validation trial is necessary to confirm that the weight, age, and estimated glomerular filtration rate based dosing regimen is able to achieve digoxin exposures consistent with the package insert recommendations.

Rationale for Dose Selection A population PK model of digoxin was developed in a cohort of 50 infants with single ventricle CHD treated with digoxin after S1P but prior to S2P. A 2 compartment model with transit compartment absorption best described the digoxin disposition in this population. Body weight and estimated glomerular filtration rate were covariates retained in the model, The model was applied to dosing simulations targeting a Cmin,ss of 0.5 - 2 ng/mL, as recommended by the digoxin package insert. Doses recommended by the model are lower than doses recommended by the current digoxin package insert, and lower that the doses received in the PTN DGX01 trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of single ventricle congenital heart disease
2. Status post-surgical or hybrid stage 1 palliation but prior to surgical stage 2 palliation
3. Age ≤ 30 days of life at time of stage 1 palliation
4. Age < 6 months at time of enrollment
5. Require treatment with enteral digoxin per their treating medical provider
6. Informed consent obtained from parent(s) or legal guardian(s)

Exclusion Criteria:

1. Gestational age at birth <35 weeks
2. Serum creatinine > 2 mg/dL at enrollment
3. Diagnosis of second degree or higher atrioventricular conduction block at enrollment
4. Diagnosis of clinically significant sinus bradycardia requiring intervention at enrollment
5. Known hypersensitivity to digoxin or other forms of digitalis
6. Extracorporeal life support (i.e., ECMO, dialysis, ventricular assist device) at enrollment
7. Received digoxin prior to enrollment
8. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 30 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Digoxin plasma concentration | End of study, up to 180 Days
  Plasma concentrations of digoxin over time measured using a validated bioanalytical assay at a central laboratory to calculate clearance and area under the curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, MD, Principal Investigator — Duke Clinical Research Institute
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No